CLINICAL TRIAL: NCT06359652
Title: Get Fit for Function Pilot Study
Brief Title: Get Fit for Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB24-0421
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Thoracic; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Prehabilitation Program Participant (Other)
  Interventions: Device: Prehabilitation Program (Apple Watch Series 6 with exercise flipbook)

INTERVENTIONS:
Device: Prehabilitation Program (Apple Watch Series 6 with exercise flipbook) — We will evaluate whether use of a personal device (the Apple Watch) could help medical professionals assess patients' pre-surgery prehab state. It will also assess whether patients are willing to use a personal device and engage in prehab exercise and whether the device can enhance prehab uptake. The intervention is to also offer patients the Exercise Flipbook, to send them a reminder to exercise and to send them notifications to track their exercise.

SUMMARY:
The purpose of this study will be to implement and evaluate a prehab program for pre-frail and frail adults who need to undergo thoracic surgery. The study team hypothesizes using an implementation framework will increase the reach, effectiveness, adoption, and implementation of the prehab program.

DETAILED DESCRIPTION:
Approximately 70% of thoracic surgery patients are pre-frail or frail, characterized by reduced strength, endurance, and physiologic function. Frailty is associated with poor perioperative outcomes, including increased complications, length of stay, post-discharge institutionalization, healthcare costs, and mortality. As a result, surgical and geriatric clinical societies now recommend including a frailty assessment in older adult pre-operative surgical evaluations. To mitigate the risks associated with frailty, prehabilitation (prehab) has been included as a component of the American College of Surgeons "Strong for Surgery" quality initiative. Evidence-based practices to optimize preoperative health have been shown to improve physical conditioning and return to autonomy, as well as, reduce length of stay, postoperative complications, and healthcare costs. Older patients who need surgery view prehab favorably, particularly if it is home-based, recommended by a medical professional, and free. The primary objective will be to conduct a feasibility evaluation using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework. The secondary objectives will be to measure functional status and clinical outcomes longitudinally in patients undergoing prehab.

Participants will receive the prehab program from 2-12 weeks prior to undergoing elective inpatient thoracic surgery. Participants will complete surveys at 2-3 weeks, 2 months, 3-4 months, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, of any racial or ethnic origin
* Will be undergoing elective thoracic surgery lung resection using thoracic approach (thoracotomy, Video-assisted thoracoscopic surgery (VATS), Robotic-Assisted Thoracic Surgery (RATS)
* Able to complete baseline evaluations at time of enrollment

Exclusion Criteria:

* Unable to give informed consent
* Unable to read/speak English
* Age <17

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
The change of functional status using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework for implementation evaluation. | At Visit 1 two to twelve weeks prior to undergoing elective inpatient thoracic surgery until post-operative Follow-up Visit up to 6 months.

SECONDARY OUTCOMES:
Number of Participants with Postoperative Complications | From Visit 2 at the time of operation until post-operative Follow-up Visit up to 6 months.
Number of Participants length of hospital stay post-operative. | From Visit 2 at the time of operation until day of discharge.
Number of Participants discharge to not-home post-operative. | From Visit 2 at the time of operation until Visit 3 for post operative clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Madariaga, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States